CLINICAL TRIAL: NCT03121846
Title: Mesylate Apatinib for Stage Ⅳ Soft Tissue Sarcoma Patients After Failure of Traditional Chemotherapy: Prospective, Open-label, Single-Arm, Multi-center Phase II Clinical Trial
Brief Title: Mesylate Apatinib for Stage Ⅳ STS After Failure of Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Gansu Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S201602
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-03

CONDITIONS: Soft Tissue Sarcoma, Adult, Stage II
Keywords: Apatinib; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib group (Experimental): apatinib 500mg po qd, 28 days for a cycle.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity.
  Other Names: Apatinib Mesylate Tablets

SUMMARY:
This is a Prospective, Open-label, Single-Arm, Multi-center phase II clinical trial evaluating the efficacy and safety of Apatinib for Chemotherapy Failure Ⅳ Stage Soft Tissue Sarcoma.

DETAILED DESCRIPTION:
The prognosis of sarcoma patients in stage IV is poor. For STS, the response rate of chemotherapy is only 20-35% and the median survival time is about 12 months. The 5 year survival rate is lower than 10% reported in several large-scale studies. Although chemotherapy plays a major role in the treatment of advanced STS, the classic chemotherapy agents are not curative. Combination chemotherapy or dose-dense regimens have largely failed to improve the response rates. Long-term using of cytotoxic drugs increased the risk of toxicity in patients. Apatinib is a small molecular inhibitor of Vascular Epithelial Growth Factor Receptor-2 (VEGFR-2). It has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance. However, the clinical application of apatinib in STS is still lack of evidence-based medicine. And this clinical trial is designed to prospectively investigate the efficacy and safety of apatinib in stage IV sarcoma patients who failed in chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join the study, signed informed consent, good compliance;
* The pathology was diagnosed as stage Ⅳ soft tissue sarcoma patients, clinical staging using the American Cancer Research Joint Committee (AJCC) TNM staging criteria. According to CT or MRI at least one measurable lesion;
* At least one chemotherapy regimen (containing anthracycline) was treated and evaluated as "disease progression" in terms of the efficacy evaluation criteria of solid tumors (RECIST 1.1).
* 18 to 70 years old, PS score: 0 ~ 2; expected survival period of more than 3 months;
* The laboratory check meets the following criteria:
* Blood routine examination: HB ≥ 100g / L (14 days without blood transfusion); ANC ≥ 1.5 × 109 / L; PLT ≥ 80 × 109 / L
* Biochemical tests: serum creatinine Cr ≤ normal upper limit (ULN), bilirubin BIL ≤ normal upper limit (ULN), ALT, AST ≤ 1.5 × normal upper limit (ULN), for liver metastases ≤ 5 × normal upper limit (ULN); fasting triglyceride ≤ 3.0mmol / L, fasting cholesterol ≤ 7.75mmol / L;
* Doppler ultrasonography: left ventricular ejection fraction (LVEF) ≥ normal low (50%).
* Women should agree that contraceptive measures (such as IUDs, contraceptives or condoms) must be used within six months of the study period and after the end of the study; serum or urine pregnancy studies were negative for 7 days prior to study , and must be non-lactating patients; men should agree that contraceptive measures must be used within six months of the study period and after the end of the study period.

Exclusion Criteria:

* Patients who have received antiangiogenic therapy or other targeted treatment for no more than 3 months, such as Endostar, Erlotinib, Sunitinib, Sorafenib, Avastin, Imatinib, Famitinib, Pazopanib and other drugs.
* Past or concurrent with other malignancies, except for cured skin basal cell carcinoma and cervical in situ cancer;
* Participated in other drug clinical researchers within four weeks;
* Previously received anticancer treatment patients with NCI CTC AE grade> 1 grade toxicity;
* Have a variety of factors that affect oral medication (such as can not swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.)
* Known brain metastases, spinal cord compression, cancerous meningitis, or screening when the CT or MRI examination found that the brain or pia mater disease;
* Patients with any severe and / or uncontrolled disease, for example:
* Unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months prior to randomization, severe uncontrollable arrhythmia; poor blood pressure control (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg )patient;
* Active or uncontrollable serious infection;
* Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;
* Poor control of diabetes (fasting blood glucose (FBG)> 10mmol / L);
* Urinary routine urinary protein ≥ ++, and confirmed 24 hours urine protein> 1.0 g;
* Long untreated wound or fracture;
* Patients with bleeding tendency (such as active gastrointestinal ulcers) or treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or analogues;
* Interventional venous thrombosis events such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism before the first medication.
* Have a history of psychiatric abuse and can not quit or have mental disorders;
* Have a history of immunodeficiency, including HIV testing positive or other acquired, congenital immune deficiency disease, or a history of organ transplantation;
* According to the researcher's judgment, there are serious illnesses that compromise the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Disease control rate(DCR） | 2 year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Objective tumor response rate(ORR) | 2 year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Overall survival(OS) | 3 year
  OS is defined as the length of time from random assignment to death or to last contact.
Adverse Events(AEs) | 2 year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jilong Yang, M.D., Ph.D., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital & Institute, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No